CLINICAL TRIAL: NCT05528510
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Guselkumab Subcutaneous Induction Therapy in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Guselkumab Therapy in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: ASTRO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109228; CNTO1959UCO3004 (Other: Janssen Research & Development, LLC); 2022-000365-41 (EudraCT Number); 2023-504719-34-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-08-19; First posted 2022-09-06 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Colitis, Ulcerative
Keywords: Guselkumab; Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Guselkumab (Experimental): Participants will receive guselkumab (Dose 1) subcutaneous (SC) injection followed by guselkumab (Dose 2) SC injection.
  Interventions: Drug: Guselkumab Dose 1; Drug: Guselkumab Dose 2
- Group 2: Guselkumab (Experimental): Participants will receive guselkumab (Dose 1) SC injection followed by guselkumab (Dose 3) SC injection.
  Interventions: Drug: Guselkumab Dose 1; Drug: Guselkumab Dose 3
- Group 3: Placebo (Placebo Comparator): Participants will receive matching placebo SC injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Guselkumab Dose 1 — Guselkumab (Dose 1) will be administered as SC injection.
  Arms: Group 1: Guselkumab; Group 2: Guselkumab
Drug: Guselkumab Dose 2 — Guselkumab (Dose 2) will be administered as SC injection.
  Arms: Group 1: Guselkumab
Drug: Guselkumab Dose 3 — Guselkumab (Dose 3) will be administered as SC injection.
  Arms: Group 2: Guselkumab
Other: Placebo — Placebo will be administered as SC injection.
  Arms: Group 3: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, including clinical remission of guselkumab subcutaneous (SC) induction compared to placebo in participants with moderately to severely active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* 18 years of age or older
* Documented diagnosis of ulcerative colitis (UC) at least 12 weeks prior to screening
* Moderately to severely active UC as per the modified Mayo score
* Demonstrated inadequate response to or intolerance of conventional therapy and/or advanced therapy as defined in the protocol

Exclusion Criteria:

* Diagnosis of indeterminate colitis, microscopic colitis, ischemic colitis, or Crohn's disease
* Surgery within 8 weeks before screening or planned surgery during the study that may confound the evaluation of benefit from study intervention
* Receiving prohibited medications and treatments
* UC limited to the rectum only
* Active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) corona virus disease (COVID-19) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2028-10-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (235):
- United States (32):
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Om Research LLC, Apple Valley, California
  - Om Research LLC, Lancaster, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Gastro Florida, Clearwater, Florida
  - I.H.S. Health. LLC, Kissimmee, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Theia Clincial Research, LLC, Temple Terrace, Florida
  - Digestive Healthcare of Georgia, P.C, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterology Associates of Central GA, Macon, Georgia
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Smart Medical Research, Hollis, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio LLC, Westlake, Ohio
  - Allegheny General Hospital of Research, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, Uniontown, Pennsylvania
  - Gastroenterology Associates of Orangeburg, SC, Orangeburg, South Carolina
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - UT Health Science Center at San Antonio, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Victoria Gastroenterology, Victoria, Texas
  - Care Access Research, Ogden, Ogden, Utah
  - Gastroenterology Associates, Salt Lake City, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
- Argentina (8):
  - Cer Instituto Medico, Buenos Aires
  - Hospital General de Agudos José Maria Ramos Mejía, Buenos Aires
  - Clinica Adventista Belgrano, Ciudad de Buenos Aires
  - Sanatorio Duarte Quiroz, Córdoba
  - Hospital Privado Universitario De Cordoba, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Hospital Provincial del Centenario, Rosario
- Australia (9):
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Health, Clayton
  - Royal Brisbane and Women's Hospital, Herston
  - Fiona Stanley Hospital, Murdoch
  - Royal Melbourne Hospital, Parkville
  - IBD Clinical Trials Mater Research, South Brisbane
  - The Queen Elizabeth Hospital, Woodville South
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (3):
  - Onze -Lieve-Vrouwziekenhuis, Aalst
  - CHU Saint-Pierre, Brussels
  - AZ Delta, Roeselare
- Brazil (14):
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - L2IP Instituto de Pesquisas Clinicas, Brasília
  - Sociedade Campineira de Educacao e Instrucao Hospital e Maternidade Celso Pierro, Campinas
  - CDC - Centro Digestivo de Curitiba, Curitiba
  - CECIP Jau - Centro de Estudos Clínicos do Interior Paulista Ltda, Jaú
  - Galileo Pesquisa Clinica, Juiz de Fora
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - CLIAGEN - Clinica de Atencao em Gastroenterologia Especializada e Nutricao, Salvador
  - Pesquisare Saude, Santo André
  - Kaiser Hospta, São José do Rio Preto
  - BR TRIALS Ensaios Clinicos e Consultoria Ltda, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
  - INTEGRAL Pesquisa e Ensino, Votuporanga
- Bulgaria (3):
  - Medical centre Asklepion, Sofia
  - DCC Convex EOOD, Sofia
  - Medical Center Leo Clinic EOOD, Targovishte
- Canada (3):
  - Fraser Clinical Trials Inc., New Westminster, British Columbia
  - Barrie GI Associates, Barrie, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
- China (25):
  - China Japan Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - West China Hospital Sichuan University, Chengdu
  - Chongqing General Hospital, Chongqing
  - First Affiliated Hospital of Gannan Medical University, Ganzhou
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - ZhuJiang Hospital of Southern Medical University, Guangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Jinhua municipal central hospital, Jinhua
  - Lanzhou University Second Hospital, Lanzhou
  - The first affiliated hospital of Henan University of science and technology, Luoyang
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Shenzhen Hospital of Southern Medical University, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Taihe Hospital, Shiyan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People s Hospital, Wuxi
  - General Hospital of Ningxia Medical Hospital, Yinchuan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
- Czechia (6):
  - Nemocnice Ceske Budejovice a s, České Budějovice
  - Gastroenterologie, s.r.o., Hradec Kralove, Hradec Kralova
  - Artroscan s r o, Ostrava
  - Synexus Czech s.r.o., Prague
  - AXON Clinical s.r.o., Prague
  - ISCARE a.s., Prague
- France (13):
  - CHRU Besancon Hopital Jean Minjoz, Besançon
  - Hopital de Bicetre, Le Kremlin-Bicêtre
  - CHRU Montpellier - Hopital Saint-Eloi, Montpellier
  - Clinique Ambroise Pare, Neuilly-sur-Seine
  - CHU de Nice Hopital de l Archet, Nice
  - Polyclinique Du Grand Sud, Nîmes
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Hospices Civils de Lyon HCL, Pierre-Bénite
  - CHU de Reims, Reims
  - Hopital d'Instruction des Armees BEGIN, Saint-Mandé
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHU Rangueil, Toulouse
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Medizinisches Versorgungszentrum (MVZ) Dachau, Dachau
  - MVZ Sanaklinikum Duisburg, Duisburg
  - Medizinische Hochschule Hannover, Hanover
  - Praxisgemeinschaft Jerichow, Jerichow
  - Staedtisches Klinikum Lueneburg, Lüneburg
- Hungary (4):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Semmelweis Egyetem AOK, Budapest
  - Vasutegeszsegugyi Nonprofit Kozhasznu Kft Debreceni Kozpont, Debrecen
- India (5):
  - Fortis Memorial Research Institute, Gurugram
  - Asian Institute Of Gastroenterology, Hyderabad
  - Kasturba Medical College Hospital, Manipal
  - P D Hinduja National Hospital and Medical Research Center, Mumbai
  - SIDS (Surat Institute of Digestive Sciences) Hospital and Research Centre, Surat
- Israel (7):
  - Ha'Emek Medical Center, Afula
  - Bnai Zion Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center - Jerusalem, ISRAEL, Jerusalem
  - Lev Talpiot Clinic, Jerusalem
  - Galilee Medical Center, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
- Japan (32):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Ginza central clinic, Chūōku
  - Sai Gastroenterology Proctology, Fujiidera-shi
  - Fukuoka University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Hachinohe City Hospital, Hachinohe
  - Tokai University Hachioji Hospital, Hachiōji
  - Matsuda Hospital, Hamamatsu
  - National Hospital Organization Mito Medical Center, Higashiibaraki-gun
  - Kagoshima University Hospital, Kagoshima
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Kyushu Rosai Hospital, Kitakyushu
  - Kumagaya General Hospital, Kumagaya-shi
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure
  - Tokushukai Chiba-Nishi General Hospital, Matsudo
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - Yokoyama IBD Clinic, Nagoya
  - Okayama Saiseikai General Hospital, Okayama
  - Kinshukai Infusion Clinic, Osaka
  - Japanese Red Cross Osaka Hospital, Osaka
  - Oita Red Cross Hospital, Ōita
  - Ishida Clinic of IBD and Gastroenterology, Ōita
  - Kindai University Hospital, Ōsaka-sayama
  - Dokkyo Medical University Hospital, Shimotsuga Gun
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku Ku
  - Tokyo Metropolitan Bokutoh Hospital, Sumida Ku
  - National Hospital Organization Shizuoka Medical Center, Sunto-gun
  - Juntendo University Hospital Urayasu, Urayasu
  - Kanke Gastrointestinal Clinic, Utsunomiya
  - Yokohama City University Medical Center, Yokohama
- Jordan (4):
  - The Speciality Hospital (TSH) / Advanced Clinical Center, Amman
  - Jordan University Hospital, Amman
  - Irbid Specialty Hospital, Aydoun
  - King Abdullah University Hospital, Irbid
- Malaysia (6):
  - Hospital Selayang, Batu Caves
  - Hospital Pulau Pinang, George Town
  - Hospital Sultanah Aminah, Johor Bahru
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - Hospital Tuanku Jaafar, Seremban
- Mexico (10):
  - SCIENTIA Investigacion Clinica SC, Chihuahua City
  - Clinica de Investigacion en Reumatologia y Obesidad, Guadalajara
  - Clinicos Asociados BOCM, SC, Mexico City
  - Centro de Investigacion Clinica Acelerada S.C, Mexico City
  - Hospital Médica Sur Tlalpan, Mexico City
  - Medical Care & Research SA de CV, Mérida
  - Centro Regiomontano de Estudios Clínicos Roma S.C., Monterrey
  - Fundacion Santos Y De La Garza Evia IBP, Monterrey
  - Clinical Research Institute Saltillo S.A. de C.V., Saltillo
  - Oncare, San Pedro Garza García
- New Zealand (5):
  - Hutt Hospital, Boulcott
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Auckland City Hospital, Grafton
  - Waikato Hospital, Hamilton
- Poland (15):
  - Gastromed Kralisz Romatowski Stachurska Sp. j., Bialystok
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Lukamed, Chojnice
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne Promed, Krakow
  - Zespol Poradni Specjalistycznych REUMED Filia nr 2, Lublin
  - EMC Instytut Medyczny SA PL CERTUS, Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - GASTROMED Sp. z o.o., Torun
  - Bodyclinic Sp. z o.o. sp. k, Warsaw
  - Medical Network Spolka z o.o. WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Przychodnia Vistamed, Wroclaw
  - Melita Medical Sp. z o.o., Wroclaw
  - Pro Life Medica Sp z o o ETG Zamosc, Zamość
- Slovakia (4):
  - FNsP F.D.R. Banska Bystrica, Banská Bystrica
  - Cliniq s.r.o., Bratislava
  - ENDOMED s.r.o, Košice
  - KM Management spol. s r.o., Nitra
- South Korea (11):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Chosun university hospital, Gwangju
  - Korea University Ansan Hospital, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - The Catholic university of Korea ST Vincent Hospital, Suwon
- Spain (4):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Virgen Macarena, Seville
  - Hosp. de La Marina Baixa, Villajoyosa
  - Hosp. Univ. Miguel Servet, Zaragoza
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
- Turkey (Türkiye) (3):
  - Istanbul University, Istanbul
  - Ege University Medical Faculty, Izmir
  - Mersin University Medical Faculty, Mersin

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Long M, Allegretti JR, Danese S, Germinaro M, Baker T, Alvarez Y, Kavalam M, Han C, Jorgens S, Jiang L, Zhang H, Hisamatsu T, Rubin DT, Peyrin-Biroulet L; ASTRO Study Group. Efficacy and safety of subcutaneous guselkumab induction therapy in participants with moderately to severely active ulcerative colitis (ASTRO): a double-blind, treat-through, randomised, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2026 Jan 13:S2468-1253(25)00322-X. doi: 10.1016/S2468-1253(25)00322-X. Online ahead of print. PMID 41544637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Results are currently reported up to the primary completion date (02-Apr-2024). Results of remaining duration will be posted upon study completion.
Groups:
- Placebo: Participants received placebo matching to guselkumab subcutaneous (SC) injection every 4 weeks (q4w) from Week 0 through Week 24. All participants in the placebo group who met rescue criteria at Week 16 received rescue treatment, that is, guselkumab 400 milligrams (mg) SC injection at Weeks 16, 20, and 24.
- Guselkumab 400 mg q4w - Guselkumab 100 mg q8w: Participants received guselkumab 400 mg SC injection at Weeks 0, 4, and 8 followed by guselkumab 100 mg SC injection every 8 weeks (q8w) starting from Week 16 through Week 24. Participants who met rescue criteria at Week 16 continued their assigned treatment regimen and received blinded sham rescue with matching placebo SC injections at Weeks 16, 20, and 24.
- Guselkumab 400 mg q4w - Guselkumab 200 mg q4w: Participants received guselkumab 400 mg SC injection at Weeks 0, 4, and 8 followed by guselkumab 200 mg SC injection q4w starting from Week 12 through Week 24. Participants who met rescue criteria at Week 16 continued their assigned treatment regimen and received blinded sham rescue with matching placebo SC injections at Weeks 16, 20, and 24.
Period: Overall Study
Arm/Group | Placebo | Guselkumab 400 mg q4w - Guselkumab 100 mg q8w | Guselkumab 400 mg q4w - Guselkumab 200 mg q4w
Started | 139 | 139 | 140
Participants Who Started Rescue Medication | 52 | 27 | 23
Completed | 131 | 136 | 136
Not Completed | 8 | 3 | 4
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 3
Not completed — Other | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Guselkumab 400 mg q4w - Guselkumab 100 mg q8w | Guselkumab 400 mg q4w - Guselkumab 200 mg q4w | Total
Number analyzed (Participants) | 139 | 139 | 140 | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.58) | 42.1 (14.59) | 43.6 (14.27) | 41.7 (14.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 60 | 53 | 162
  Male | 90 | 79 | 87 | 256
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 30 | 26 | 79
  Not Hispanic or Latino | 112 | 102 | 112 | 326
  Unknown or Not Reported | 4 | 7 | 2 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 0 | 4
  Asian | 40 | 41 | 40 | 121
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 6 | 6 | 13
  White | 94 | 85 | 91 | 270
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 3 | 2 | 2 | 7
AgeCategorical [Count of Participants; unit: Participants]
  Adults (18-64 years) | 131 | 123 | 131 | 385
  65 years and over | 8 | 16 | 9 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 4 | 4 | 3 | 11
  AUSTRALIA | 2 | 2 | 3 | 7
  BELGIUM | 0 | 2 | 0 | 2
  BRAZIL | 17 | 18 | 19 | 54
  BULGARIA | 1 | 2 | 1 | 4
  CANADA | 1 | 0 | 0 | 1
  CHINA | 19 | 12 | 16 | 47
  CZECH REPUBLIC | 4 | 5 | 3 | 12
  FRANCE | 3 | 6 | 3 | 12
  GERMANY | 2 | 1 | 2 | 5
  HUNGARY | 3 | 1 | 4 | 8
  INDIA | 3 | 2 | 8 | 13
  ISRAEL | 2 | 2 | 2 | 6
  JAPAN | 7 | 15 | 10 | 32
  JORDAN | 9 | 6 | 6 | 21
  MALAYSIA | 2 | 3 | 2 | 7
  MEXICO | 1 | 5 | 6 | 12
  NEW ZEALAND | 3 | 1 | 0 | 4
  POLAND | 31 | 28 | 34 | 93
  SLOVAKIA | 2 | 0 | 0 | 2
  SOUTH KOREA | 7 | 6 | 2 | 15
  SPAIN | 5 | 1 | 0 | 6
  TAIWAN | 0 | 3 | 1 | 4
  TURKEY | 1 | 4 | 2 | 7
  UNITED STATES | 10 | 10 | 13 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Clinical Remission at Week 12
Description: Percentage of participants in clinical remission at Week 12 was reported. Clinical remission is defined as a Mayo stool frequency subscore of 0 or 1 and not increased from baseline, a Mayo rectal bleeding subscore of 0, and a Mayo endoscopy subscore of 0, or 1 with no friability present on the endoscopy. Mayo stool frequency subscore was determined on the average number of stools more than normal in 24 hours, score ranged from 0 (normal number of stools) to 3 (5 or more stools more than normal), higher score indicated more severity. Mayo rectal bleeding subscore ranged from 0 (no blood seen) to 3 (blood alone passed), higher score indicated more severity. Mayo endoscopy subscore ranged from 0 (normal or inactive disease) to 3 (severe disease), higher score indicated more severity.
Time Frame: Week 12
Population: Full analysis set (FAS) included all randomized participants who received at least 1 (partial or complete) dose of study intervention. As planned, combined data of guselkumab 400 mg SC induction dose group (that is, participants from guselkumab groups: 100 mg SC q8w and 200 mg SC q4w that received same induction dose of Guselkumab 400 mg SC q4w at Weeks 0, 4, and 8) is reported.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Combined Guselkumab 400 mg: Participants received guselkumab 400 mg SC injection at Weeks 0, 4, and 8. This arm includes all participants that received guselkumab 400 mg induction dose.
Arm/Group | Placebo | Combined Guselkumab 400 mg
Number analyzed (Participants) | 139 | 279
Percentage of participants | 6.5 [2.4 to 10.6] | 27.6 [22.4 to 32.8]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.001, Mantel Haenszel; Stratification was by Androgen Deprivation Therapy for Intermediate-Risk status (Yes/No) and Mayo endoscopy subscore at baseline(moderate or severe); Adjusted Treatment Difference = 21.1, 95% CI 2-sided [14.5 to 27.6]

2. Secondary Outcome: Percentage of Participants in Symptomatic Remission at Week 12
Description: Percentage of participants in symptomatic remission at Week 12 was reported. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and not increased from baseline, and a rectal bleeding subscore of 0. Mayo stool frequency subscore was determined on the average number of stools more than normal in 24 hours, score ranged from 0 (normal number of stools) to 3 (5 or more stools more than normal), higher score indicated more severity. Mayo rectal bleeding subscore ranged from 0 (no blood seen) to 3 (blood alone passed), higher score indicated more severity.
Time Frame: Week 12
Population: FAS included all randomized participants who received at least 1 (partial or complete) dose of study intervention. As planned, combined data of guselkumab 400 mg SC induction dose group (that is, participants from guselkumab groups: 100 mg SC q8w and 200 mg SC q4w that received same induction dose of Guselkumab 400 mg SC q4w at Weeks 0, 4, and 8) is reported.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Combined Guselkumab 400 mg
Number analyzed (Participants) | 139 | 279
Percentage of participants | 20.9 [14.1 to 27.6] | 51.3 [45.4 to 57.1]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 30.4, 95% CI 2-sided [21.6 to 39.2]

3. Secondary Outcome: Percentage of Participants With Endoscopic Improvement at Week 12
Description: Percentage of participants with endoscopic improvement at Week 12 was reported. Endoscopic improvement is defined as an endoscopy subscore of 0, or 1 with no friability present on the endoscopy. Mayo endoscopy subscore ranged from 0 (normal or inactive disease) to 3 (severe disease), higher score indicated more severity.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Combined Guselkumab 400 mg
Number analyzed (Participants) | 139 | 279
Percentage of participants | 12.9 [7.4 to 18.5] | 37.3 [31.6 to 42.9]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 24.3, 95% CI 2-sided [16.6 to 31.9]

4. Secondary Outcome: Percentage of Participants in Clinical Response at Week 12
Description: Percentage of participants in clinical response at Week 12 was reported. Clinical response is defined as a decrease from baseline in the modified Mayo score by greater than or equal to (>=) 30 percent (%) and >=2 points, with either a >=1-point decrease from baseline in the rectal bleeding subscore or a rectal bleeding subscore of 0 or 1. The modified Mayo scores consisted of 3 subscores: stool frequency, rectal bleeding and endoscopic subscore, each subscore graded from 0 (normal) to 3 (severe) with higher scores indicating more severe disease. These individual subscores were summed up to give a total modified Mayo score range of 0 (normal) to 9 (severe disease), where higher scores indicated more severe disease activity.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Combined Guselkumab 400 mg
Number analyzed (Participants) | 139 | 279
Percentage of participants | 34.5 [26.6 to 42.4] | 65.6 [60.0 to 71.2]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 31, 95% CI 2-sided [21.6 to 40.5]

5. Secondary Outcome: Percentage of Participants With Histologic-endoscopic Mucosal Improvement at Week 12
Description: Percentage of participants with histologic-endoscopic mucosal improvement at Week 12 was reported. Histologic-endoscopic mucosal improvement is defined as achieving a combination of histologic improvement and endoscopic improvement. Histologic improvement is defined as neutrophil infiltration in less than (<) 5% of crypts, no crypt destruction, and no erosions, ulcerations or granulation tissue according to the Geboes grading system. Endoscopic improvement is defined as an endoscopy subscore of 0, or 1 with no friability present on the endoscopy. Mayo endoscopy subscore ranged from 0 (normal or inactive disease) to 3 (severe disease), higher score indicated more severity.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Combined Guselkumab 400 mg
Number analyzed (Participants) | 139 | 279
Percentage of participants | 10.8 [5.6 to 15.9] | 30.5 [25.1 to 35.9]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 19.6, 95% CI 2-sided [12.4 to 26.9]

6. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 24
Description: Percentage of participants in clinical remission at Week 24 was reported. Clinical remission is defined as a stool frequency subscore of 0 or 1 and not increased from baseline, a rectal bleeding subscore of 0, and an endoscopy subscore of 0, or 1 with no friability present on the endoscopy. Mayo stool frequency subscore was determined on the average number of stools more than normal in 24 hours, score ranged from 0 (normal number of stools) to 3 (5 or more stools more than normal), higher score indicated more severity. Mayo rectal bleeding subscore ranged from 0 (no blood seen) to 3 (blood alone passed), higher score indicated more severity. Mayo endoscopy subscore ranged from 0 (normal or inactive disease) to 3 (severe disease), higher score indicated more severity.
Time Frame: Week 24
Population: FAS included all randomized participants who received at least 1 (partial or complete) dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Guselkumab 400 mg q4w - Guselkumab 100 mg q8w | Guselkumab 400 mg q4w - Guselkumab 200 mg q4w
Number analyzed (Participants) | 139 | 139 | 140
Percentage of participants | 9.4 [4.5 to 14.2] | 35.3 [27.3 to 43.2] | 36.4 [28.5 to 44.4]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 400 mg q4w - Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 25.9, 95% CI 2-sided [16.7 to 35.1]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 400 mg q4w - Guselkumab 200 mg q4w; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 27, 95% CI 2-sided [17.9 to 36.2]

7. Secondary Outcome: Percentage of Participants in Symptomatic Remission at Week 24
Description: Percentage of participants in symptomatic remission at Week 24 was reported. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and not increased from baseline, and a rectal bleeding subscore of 0. Mayo stool frequency subscore was determined on the average number of stools more than normal in 24 hours, score ranged from 0 (normal number of stools) to 3 (5 or more stools more than normal), higher score indicated more severity. Mayo rectal bleeding subscore ranged from 0 (no blood seen) to 3 (blood alone passed), higher score indicated more severity.
Time Frame: Week 24
Population: FAS included all randomized participants who received at least 1 (partial or complete) dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Guselkumab 400 mg q4w - Guselkumab 100 mg q8w | Guselkumab 400 mg q4w - Guselkumab 200 mg q4w
Number analyzed (Participants) | 139 | 139 | 140
Percentage of participants | 25.2 [18.0 to 32.4] | 54.7 [46.4 to 63.0] | 50.0 [41.7 to 58.3]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 400 mg q4w - Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 29.5, 95% CI 2-sided [18.5 to 40.5]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 400 mg q4w - Guselkumab 200 mg q4w; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 24.8, 95% CI 2-sided [14.3 to 35.3]

8. Secondary Outcome: Percentage of Participants With Endoscopic Improvement at Week 24
Description: Percentage of participants with endoscopic improvement at Week 24 was reported. Endoscopic improvement is defined as an endoscopy subscore of 0, or 1 with no friability present on the endoscopy. Mayo endoscopy subscore ranged from 0 (normal or inactive disease) to 3 (severe disease), higher score indicated more severity.
Time Frame: Week 24
Population: FAS included all randomized participants who received at least 1 (partial or complete) dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Guselkumab 400 mg q4w - Guselkumab 100 mg q8w | Guselkumab 400 mg q4w - Guselkumab 200 mg q4w
Number analyzed (Participants) | 139 | 139 | 140
Percentage of participants | 12.2 [6.8 to 17.7] | 40.3 [32.1 to 48.4] | 45.0 [36.8 to 53.2]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 400 mg q4w - Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 28.1, 95% CI 2-sided [18.5 to 37.6]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 400 mg q4w - Guselkumab 200 mg q4w; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 32.7, 95% CI 2-sided [23.1 to 42.3]

9. Secondary Outcome: Percentage of Participants in Clinical Response at Week 24
Description: Percentage of participants in clinical response at Week 24 was reported. Clinical response is defined as a decrease from baseline in the modified Mayo score by >= 30% and >=2 points, with either a >=1-point decrease from baseline in the rectal bleeding subscore or a rectal bleeding subscore of 0 or 1. The modified Mayo scores consisted of 3 subscores: stool frequency, rectal bleeding and endoscopic subscore, each subscore graded from 0 (normal) to 3 (severe) with higher scores indicating more severe disease. These individual subscores were summed up to give a total modified Mayo score range of 0 (normal) to 9 (severe disease), where higher scores indicated more severe disease activity.
Time Frame: Week 24
Population: FAS included all randomized participants who received at least 1 (partial or complete) dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Guselkumab 400 mg q4w - Guselkumab 100 mg q8w | Guselkumab 400 mg q4w - Guselkumab 200 mg q4w
Number analyzed (Participants) | 139 | 139 | 140
Percentage of participants | 30.9 [23.3 to 38.6] | 63.3 [55.3 to 71.3] | 61.4 [53.4 to 69.5]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 400 mg q4w - Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 32.4, 95% CI 2-sided [21.3 to 43.4]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 400 mg q4w - Guselkumab 200 mg q4w; Test type: Superiority; p < 0.001, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Adjusted Treatment Difference = 30.5, 95% CI 2-sided [20.0 to 41.0]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From screening (-8 weeks) up to Week 24; Serious adverse events (SAEs) and Other AEs: From Week 0 up to Week 24
Description: Safety analysis set included all randomized participants who received at least 1 (partial or complete) dose of study intervention. As planned, safety data were analyzed per intervention through Week 24.
Groups:
- Placebo (Before Rescue Medication): Participants received placebo matching to guselkumab subcutaneous (SC) injection every 4 weeks (q4w) from Week 0 through Week 24. This arm includes data of all placebo participants excluding data after a participant was rescued with guselkumab.
- Placebo - Guselkumab (After Rescue Medication): All participants in the placebo group who met rescue criteria at Week 16 received rescue treatment that is guselkumab 400 milligrams (mg) mg SC injection at Weeks 16, 20, and 24. Rescue Criteria: No improvement (no decrease) in Mayo endoscopy subscore at Week 12 as obtained during central review, when compared with baseline and a less than (<) 2 point improvement (<2 point decrease) in partial Mayo score at Weeks 12 and 16, when compared with baseline. This arm includes data occurred after a participant crossed over to guselkumab.
Arm/Group | Placebo (Before Rescue Medication) | Placebo - Guselkumab (After Rescue Medication) | Guselkumab 400 mg q4w - Guselkumab 100 mg q8w | Guselkumab 400 mg q4w - Guselkumab 200 mg q4w
All-Cause Mortality (participants affected / at risk) | 1/139 | 0/52 | 0/139 | 0/140
Serious Adverse Events (participants affected / at risk) | 17/139 | 1/52 | 5/139 | 6/140
Other Adverse Events (participants affected / at risk) | 48/139 | 5/52 | 47/139 | 39/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Before Rescue Medication) (N=139) | Placebo - Guselkumab (After Rescue Medication) (N=52) | Guselkumab 400 mg q4w - Guselkumab 100 mg q8w (N=139) | Guselkumab 400 mg q4w - Guselkumab 200 mg q4w (N=140)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 11 | 1 | 2 | 2
Colon Dysplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Pilonidal Disease (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 0 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Before Rescue Medication) (N=139) | Placebo - Guselkumab (After Rescue Medication) (N=52) | Guselkumab 400 mg q4w - Guselkumab 100 mg q8w (N=139) | Guselkumab 400 mg q4w - Guselkumab 200 mg q4w (N=140)
Anaemia (Blood and lymphatic system disorders) | 8 | 2 | 5 | 5
Abdominal Pain (Gastrointestinal disorders) | 5 | 0 | 2 | 2
Colitis Ulcerative (Gastrointestinal disorders) | 19 | 1 | 12 | 7
Injection Site Erythema (General disorders) | 1 | 1 | 4 | 6
Covid-19 (Infections and infestations) | 5 | 1 | 5 | 2
Nasopharyngitis (Infections and infestations) | 8 | 0 | 5 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 0 | 10 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 11 | 7
Headache (Nervous system disorders) | 3 | 0 | 7 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study site and investigator shall not publish study results except as required by law or as specified in a separate, written agreement between the sponsor and the study site or investigator. Sponsor will register the study and publish the study results in compliance with applicable law and may register the study or publish study results when not required.

DOCUMENTS (2):
  • Study Protocol (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT05528510/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT05528510/SAP_001.pdf